CLINICAL TRIAL: NCT03655717
Title: Using Imaging to Assess Effects of THC on Brain Activity
Acronym: fNIRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, A. Eden Evins, Director, Center for Addiction Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2015P001516; R42DA043977 (NIH)
Record Dates: First submitted 2018-07-20; First posted 2018-08-31 (Actual); Results first posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Intoxication Alcohol; Intoxication THC; Intoxication Combined Alcohol THC
Keywords: fNIRS; THC; Intoxication
MeSH Terms: conditions — Alcoholic Intoxication | interventions — Dronabinol; Ethanol

STUDY DESIGN:
Intervention Model Description: In Phase 2A, a double-blind placebo-controlled, random order cross-over study of single dose dronabinol, participants received dronabinol or identical placebo on two separate study visits in randomized order.
  In Phase 2B, a randomized, double-blind, 4-treatment, 4-period, crossover study with THC or placebo administration and ethanol or placebo administration, participants were randomly assigned to 1 of 24 sequences of each of the following treatments: placebo dronabinol and placebo ethanol, placebo dronabinol and ethanol, dronabinol and placebo ethanol, and dronabinol and ethanol.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects will be randomly assigned to one of the possible orders according to a randomization schedule generated by the study staff using a random number generator and computer program. The Massachusetts General Hospital (MGH) research pharmacy will generate a blinded randomization code for order of dosing and will dispense blinded drug in the dose ordered and identical placebo for use on separate study days. Ethanol or placebo drink will be prepared by a member of the research unit staff not otherwise associated with study visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 2A (Experimental): In a double-blind placebo-controlled, random order cross-over study of single dose dronabinol, participants received dronabinol or identical placebo on two separate study visits in randomized order.
  Interventions: Drug: Dronabinol; Drug: Placebo dronabinol
- Phase 2B (Experimental): In a randomized, double-blind, 4-treatment, 4-period, crossover study with THC or placebo administration and ethanol or placebo administration, participants were randomly assigned to 1 of 4 sequences and received each of the following treatments: placebo dronabinol + placebo ethanol, placebo dronabinol + ethanol, dronabinol + placebo ethanol, & dronabinol + ethanol.
  Interventions: Drug: Dronabinol; Drug: Ethanol; Drug: Placebo dronabinol; Drug: Placebo ethanol

INTERVENTIONS:
Drug: Dronabinol — Dronabinol at physician determined doses of 10-80mg designed to produce intoxication.
  Other Names: oral THC
Drug: Ethanol — Oral Ethanol, dosed to obtain a breath alcohol concentration (BrAC) of approximately 0.05 BrAC (equal to 1-2 standard drinks).
  Other Names: oral ethanol
  Arms: Phase 2B
Drug: Placebo dronabinol — Identical in appearance to active dronabinol (overencapsulation of both active and placebo dronabinol)
  Other Names: placebo oral THC
Drug: Placebo ethanol — Placebo ethanol will consist of diet soda used in the active ethanol condition with 0.25ml ethanol floated on top to provide the odor of ethanol and blind the study drug.
  Other Names: oral placebo ethanol
  Arms: Phase 2B

SUMMARY:
This study will assess effects of tetrahydrocannabinol (THC) and THC + alcohol in marijuana users on prefrontal brain activity, using functional near-infrared spectroscopy (fNIRS) during resting state and during memory task performance. Participants will complete fNIRS testing 120 minutes following THC or identical placebo (Phase 2A), or THC/ethanol, THC/placebo ethanol, placebo THC/ethanol, and placebo THC/placebo ethanol (Phase 2B), and oxygenated hemoglobin (HbO) concentration will be measured.

DETAILED DESCRIPTION:
This study will assess the effects of THC intoxication using dronabinol (synthetic THC) on the oxyhemoglobin (HbO) signal during resting state and task-based activation in the prefrontal cortex (PFC) and resting state connectivity, as well as on neurocognitive task performance and correlations between these measurements and clinical signs of intoxication. Participants will be 150 adults who use marijuana at least monthly (aged 18-55) will be recruited to participate in this study. Participants will be given up to 80 mg of dronabinol, an FDA-approved synthetic form of THC that is used to treat loss of appetite that causes weight loss in people with AIDS. THC is the principle psychoactive drug in marijuana. The study will be conducted in regular cannabis users who present at their first study visit with a positive urine screen for THC metabolites.

Phase 2A. Investigate the effect of THC on fNIRS brain signature and its association with self-reported intoxication, laboratory measures of impairment, and the gold-standard behavioral field test of driving impairment used by law enforcement, the primary classifier.

Phase 2B. Examine potential interaction following co-administration of THC with oral ethanol exposure in healthy volunteers. Phase II is a randomized, double-blind, placebo-controlled, 2 by 2 crossover study of effect of dronabinol, ethanol, and combined dronabinol and ethanol on brain activation and connectivity as measured by fNIRS.

ELIGIBILITY:
Inclusion Criteria General

1. Men and women aged 18-55 years, inclusive; (for Phase 2B: men and women aged 21-55 years, inclusive)
2. Competent and willing to provide written informed consent;
3. Able to communicate in English language.
4. Regular, at least monthly, marijuana use, confirmed by positive urine screen for THC

   Additional Inclusion Criteria For Phase 2B:
5. Past consumption of at least two alcoholic beverages in one occasion.
6. Past co-consumption of alcohol and THC at least once in lifetime with no serious adverse effects.
7. Weigh more than 100 lbs.

Exclusion Criteria:

General (Phase 2A, 2B 3)

1. Any unstable, serious medical illness, or cardiovascular disease or events.
2. New or unstable psychiatric symptoms, schizophrenia, or bipolar I disorder,
3. Diabetes, cirrhosis, renal failure, Hepatitis C, HIV,
4. History of syncope without an identified situational stressor, migraines >1x/month, head injury with prolonged unconsciousness (> 24 hours);
5. Allergy to sesame oil (contained in Marinol pills) or Marinol capsules
6. Daily use of benzodiazepines or barbiturates, antihistamines, atropine, scopolamine, or other strong anticholinergic agents;
7. Current pregnancy or lactation, or trying to become pregnant (confirmed by urine pregnancy test)
8. In the opinion of the investigator, not able to safely participate in this study.

   Additional Exclusion Criteria For Phase 2B:
9. Currently seeking treatment, in treatment, or in recovery from an alcohol use disorder.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 316 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Eden Evins, MD, MPH, Principal Investigator — Massachusetts General Hospital; Jodi M Gilman, PhD, Study Director — Massachusetts General Hospital
Locations (1):
- Center for Addiction Medicine, Massachusetts General Hospital, Dept. of Psychiatry, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be available

REFERENCES:
- [Derived] Berchansky M, Evins AE, Evohr B, Himmelsbach Z, Pachas GN, Karunakaran KD, Laufer Goldshtein B, Ozana N, Gilman JM. Detection of Delta9-Tetrahydrocannabinol Impairment Using Resting-State Functional Near-Infrared Spectroscopy: A Randomized Clinical Trial. JAMA Netw Open. 2026 Jan 2;9(1):e2556647. doi: 10.1001/jamanetworkopen.2025.56647. PMID 41615687
- [Derived] Karunakaran KD, Pascale M, Ozana N, Potter K, Pachas GN, Evins AE, Gilman JM. Intoxication due to Delta9-tetrahydrocannabinol is characterized by disrupted prefrontal cortex activity. Neuropsychopharmacology. 2024 Aug;49(9):1481-1490. doi: 10.1038/s41386-024-01876-5. Epub 2024 May 7. PMID 38714786
- [Derived] Gilman JM, Schmitt WA, Potter K, Kendzior B, Pachas GN, Hickey S, Makary M, Huestis MA, Evins AE. Identification of ∆9-tetrahydrocannabinol (THC) impairment using functional brain imaging. Neuropsychopharmacology. 2022 Mar;47(4):944-952. doi: 10.1038/s41386-021-01259-0. Epub 2022 Jan 8. PMID 34999737

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by study staff at the MGH Center for Addiction Medicine through advertising by email, web and bulletin board announcements posted within the local site network community.
Pre-assignment Details: A screening visit took place before randomization. After randomization, phase 2A completed two visits and phase 2B completed four visits.
  Washout achieved with at least one week between visits. Participant dropout affected by the COVID-19 pandemic.
  Due to character limit, sequences coded as follows:
  A: Placebo Dronabinol
  B: Dronabinol
  C: Placebo Dronabinol & Placebo Ethanol
  D: Dronabinol & Placebo Ethanol
  E: Placebo Dronabinol & Ethanol
  F: Dronabinol & Ethanol
Groups:
- Phase 2A: AB: Placebo then Dronabinol
  Over two visits, Phase 2A participants were assigned in a random order to a single dose of either dronabinol and placebo. Visits were approximately one week apart.
- Phase 2A: BA: Dronabinol then Placebo
- Phase 2B: CDEF: Placebo Dronabinol and Placebo Ethanol, then Dronabinol and Placebo Ethanol, then Placebo Dronabinol and Ethanol, then Dronabinol and Ethanol
  Phase 2B was a randomized, double-blind, 4-treatment, 4-period, crossover study with THC or placebo administration and ethanol or placebo administration.
  Over four visits participants were assigned in a random order to each of dronabinol and ethanol, dronabinol and placebo ethanol, placebo dronabinol and ethanol, or placebo dronabinol and placebo ethanol. Visits were approximately one week apart.
- Phase 2B: CDFE: Placebo Dronabinol and Placebo Ethanol, then Dronabinol and Placebo Ethanol, then Dronabinol and Ethanol, then Placebo Dronabinol and Ethanol
- Phase 2B: CEDF: Placebo Dronabinol and Placebo Ethanol, then Placebo Dronabinol and Ethanol, then Dronabinol and Placebo Ethanol, then Dronabinol and Ethanol
- Phase 2B: CEFD: Placebo Dronabinol and Placebo Ethanol, then Placebo Dronabinol and Ethanol, then Dronabinol and Ethanol, then Dronabinol and Placebo Ethanol
- Phase 2B: CFDE: Placebo Dronabinol and Placebo Ethanol, then Dronabinol and Ethanol, then Dronabinol and Placebo Ethanol, then Placebo Dronabinol and Ethanol
- Phase 2B: CFED: Placebo Dronabinol and Placebo Ethanol, then Dronabinol and Ethanol, then Placebo Dronabinol and Ethanol, then Dronabinol and Placebo Ethanol
- Phase 2B: DCEF: Dronabinol and Placebo Ethanol, then Placebo Dronabinol and Placebo Ethanol, then Placebo Dronabinol and Ethanol, then Dronabinol and Ethanol
- Phase 2B: DCFE: Dronabinol and Placebo Ethanol, then Placebo Dronabinol and Placebo Ethanol, then Dronabinol and Ethanol, then Placebo Dronabinol and Ethanol
- Phase 2B: DECF: Dronabinol and Placebo Ethanol, then Placebo Dronabinol and Ethanol, then Placebo Dronabinol and Placebo Ethanol, then Dronabinol and Ethanol
- Phase 2B: DEFC: Dronabinol and Placebo Ethanol, then Placebo Dronabinol and Ethanol, then Dronabinol and Ethanol, then Placebo Dronabinol and Placebo Ethanol
- Phase 2B: DFCE: Dronabinol and Placebo Ethanol, then Dronabinol and Ethanol, then Placebo Dronabinol and Placebo Ethanol, then Placebo Dronabinol and Ethanol
- Phase 2B: DFEC: Dronabinol and Placebo Ethanol, then Dronabinol and Ethanol, then Placebo Dronabinol and Ethanol, then Placebo Dronabinol and Placebo Ethanol
- Phase 2B: ECDF: Placebo Dronabinol and Ethanol, then Placebo Dronabinol and Placebo Ethanol, then Dronabinol and Placebo Ethanol, then Dronabinol and Ethanol
- Phase 2B: ECFD: Placebo Dronabinol and Ethanol, then Placebo Dronabinol and Placebo Ethanol, then Dronabinol and Ethanol, then Dronabinol and Placebo Ethanol
- Phase 2B: EDCF: Placebo Dronabinol and Ethanol, then Dronabinol and Placebo Ethanol, then Placebo Dronabinol and Placebo Ethanol, then Dronabinol and Ethanol
- Phase 2B: EDFC: Placebo Dronabinol and Ethanol, then Dronabinol and Placebo Ethanol, then Dronabinol and Ethanol, then Placebo Dronabinol and Placebo Ethanol
- Phase 2B: EFCD: Placebo Dronabinol and Ethanol, then Dronabinol and Ethanol, then Placebo Dronabinol and Placebo Ethanol, then Dronabinol and Placebo Ethanol
- Phase 2B: EFDC: Placebo Dronabinol and Ethanol, then Dronabinol and Ethanol, then Dronabinol and Placebo Ethanol, then Placebo Dronabinol and Placebo Ethanol
- Phase 2B: FCDE: Dronabinol and Ethanol, then Placebo Dronabinol and Placebo Ethanol, then Dronabinol and Placebo Ethanol, then Placebo Dronabinol and Ethanol
- Phase 2B: FCED: Dronabinol and Ethanol, then Placebo Dronabinol and Placebo Ethanol, then Placebo Dronabinol and Ethanol, then Dronabinol and Placebo Ethanol
- Phase 2B: FDCE: Dronabinol and Ethanol, then Dronabinol and Placebo Ethanol, then Placebo Dronabinol and Placebo Ethanol, then Placebo Dronabinol and Ethanol
- Phase 2B: FDEC: Dronabinol and Ethanol, then Dronabinol and Placebo Ethanol, then Placebo Dronabinol and Ethanol, then Placebo Dronabinol and Placebo Ethanol
- Phase 2B: FECD: Dronabinol and Ethanol, then Placebo Dronabinol and Ethanol, then Placebo Dronabinol and Placebo Ethanol, then Dronabinol and Placebo Ethanol
- Phase 2B: FEDC: Dronabinol and Ethanol, then Placebo Dronabinol and Ethanol, then Dronabinol and Placebo Ethanol, then Placebo Dronabinol and Placebo Ethanol
Period: Overall Study
Arm/Group | Phase 2A: AB | Phase 2A: BA | Phase 2B: CDEF | Phase 2B: CDFE | Phase 2B: CEDF | Phase 2B: CEFD | Phase 2B: CFDE | Phase 2B: CFED | Phase 2B: DCEF | Phase 2B: DCFE | Phase 2B: DECF | Phase 2B: DEFC | Phase 2B: DFCE | Phase 2B: DFEC | Phase 2B: ECDF | Phase 2B: ECFD | Phase 2B: EDCF | Phase 2B: EDFC | Phase 2B: EFCD | Phase 2B: EFDC | Phase 2B: FCDE | Phase 2B: FCED | Phase 2B: FDCE | Phase 2B: FDEC | Phase 2B: FECD | Phase 2B: FEDC
Started | 70 | 68 | 2 | 1 | 0 | 3 | 3 | 3 | 2 | 1 | 1 | 3 | 2 | 3 | 2 | 2 | 2 | 2 | 3 | 3 | 2 | 3 | 2 | 4 | 1 | 2
Completed | 60 | 56 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 0 | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 2 | 0 | 2
Not Completed | 10 | 12 | 1 | 1 | 0 | 2 | 3 | 1 | 2 | 1 | 0 | 2 | 0 | 3 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 8 | 1 | 0 | 0 | 1 | 3 | 1 | 2 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 0
Not completed — Physician Decision | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 3 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 2A - Total Sample: In a double-blind placebo-controlled, random order cross-over study of single dose dronabinol, participants received dronabinol or identical placebo on two separate study visits in randomized order.
- Phase 2B - Total Sample: In a randomized, double-blind, 4-treatment, 4-period, crossover study with THC or placebo administration and ethanol or placebo administration, participants were randomly assigned to 1 of 4 sequences and received each of the following treatments: placebo dronabinol + placebo ethanol, placebo dronabinol + ethanol, dronabinol + placebo ethanol, & dronabinol + ethanol.
- Total: Total of all reporting groups
Arm/Group | Phase 2A - Total Sample | Phase 2B - Total Sample | Total
Number analyzed (Participants) | 138 | 52 | 190
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 138 | 52 | 190
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.9 (6.49) | 25.6 (5.16) | 25.1 (6.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 27 | 94
  Male | 71 | 25 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 10 | 38
  Not Hispanic or Latino | 107 | 41 | 148
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 11 | 2 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 6 | 22
  White | 93 | 36 | 129
  More than one race | 12 | 4 | 16
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 138 | 52 | 190

OUTCOME MEASURES:

1. Primary Outcome: Change in Concentration of Oxygenated Hemoglobin Between Pre-drug and Post-drug Scans of Patients Completing the N-back Task.
Description: Subjects completed the N-back task before and after receiving a combination of active dronabinol or placebo dronabinol and active ethanol or placebo ethanol. During the task, the fNIRS device was used to capture change in concentration of oxygenated hemoglobin to assess prefrontal brain activity.
  Outcomes reflect average change from baseline in HbO concentration over pre-dose scan and average change from baseline in HbO concentration over post-dose scan (expected peak intoxication).
Time Frame: The first Nback scan session was run before dosing (t ≈ -35min). Drug was administered (t = 0min). The second Nback scan session was run at the time of expected peak pharmacokinetic effect (t ≈ 100min). Each scan session was six minutes in duration.
Population: Note: The Participant Flow lists Phase 2A by randomization sequence (recommended for crossover studies).
  Phase 2A: Includes participants that completed scans after receiving dronabinol (119 subjects) and after placebo (115 subjects) Phase 2B: Incudes participants that completed scans after receiving dronabinol + ethanol (30 subjects), dronabinol + placebo ethanol (31 subjects), placebo dronabinol + ethanol (28 subjects) and placebo dronabinol + placebo ethanol (34 subjects)
Measure: Mean (Standard Deviation); unit: Δ mol/L
Groups:
- Phase 2A: Dronabinol Only: This group includes the Phase 2A visit at which dronabinol was administered.
  Phase 2A was a double-blind placebo-controlled, random order cross-over study in which participants received dronabinol or identical placebo on two separate study visits, one week apart.
- Phase 2A: Placebo Dronabinol Only: This group includes the Phase 2A visit at which placebo dronabinol was administered.
  Phase 2A was a double-blind placebo-controlled, random order cross-over study in which participants received dronabinol or identical placebo on two separate study visits, one week apart.
- Phase 2B: Dronabinol and Ethanol: Phase 2B was a randomized, double-blind, 4-treatment, 4-period, crossover study with THC or placebo administration and ethanol or placebo administration.
  Over four visits participants were assigned in a random order to each of dronabinol and ethanol, dronabinol and placebo ethanol, placebo dronabinol and ethanol, or placebo dronabinol and placebo ethanol. Visits were approximately one week apart.
  At this visit, participants received dronabinol and ethanol.
- Phase 2B: Dronabinol and Placebo Ethanol: Phase 2B was a randomized, double-blind, 4-treatment, 4-period, crossover study with THC or placebo administration and ethanol or placebo administration.
  Over four visits participants were assigned in a random order to each of dronabinol and ethanol, dronabinol and placebo ethanol, placebo dronabinol and ethanol, or placebo dronabinol and placebo ethanol. Visits were approximately one week apart.
  At this visit, participants received dronabinol and placebo ethanol.
- Phase 2B: Placebo Dronabinol and Ethanol: Phase 2B was a randomized, double-blind, 4-treatment, 4-period, crossover study with THC or placebo administration and ethanol or placebo administration.
  Over four visits participants were assigned in a random order to each of dronabinol and ethanol, dronabinol and placebo ethanol, placebo dronabinol and ethanol, or placebo dronabinol and placebo ethanol. Visits were approximately one week apart.
  At this visit, participants received placebo dronabinol and ethanol.
- Phase 2B: Placebo Dronabinol and Placebo Ethanol: Phase 2B was a randomized, double-blind, 4-treatment, 4-period, crossover study with THC or placebo administration and ethanol or placebo administration.
  Over four visits participants were assigned in a random order to each of dronabinol and ethanol, dronabinol and placebo ethanol, placebo dronabinol and ethanol, or placebo dronabinol and placebo ethanol. Visits were approximately one week apart.
  At this visit, participants received placebo dronabinol and placebo ethanol.
Arm/Group | Phase 2A: Dronabinol Only | Phase 2A: Placebo Dronabinol Only | Phase 2B: Dronabinol and Ethanol | Phase 2B: Dronabinol and Placebo Ethanol | Phase 2B: Placebo Dronabinol and Ethanol | Phase 2B: Placebo Dronabinol and Placebo Ethanol
Number analyzed (Participants) | 119 | 115 | 30 | 31 | 28 | 34
Δ mol/L
  Predose | 0.00000000042 (0.00000011109) | -0.00000000126 (0.00000012928) | -0.00000000271 (0.00000015932) | -0.00000000114 (0.00000015048) | -0.00000000151 (0.00000009318) | -0.00000000219 (0.00000012507)
  Peak | 0.00000000013 (0.00000010190) | 0.00000000029 (0.00000012394) | -0.00000000041 (0.00000010552) | -0.00000000020 (0.00000012457) | -0.00000000018 (0.00000009089) | 0.00000000070 (0.00000011546)
Statistical Analysis 1: Comparison: Phase 2A: Dronabinol Only vs Phase 2A: Placebo Dronabinol Only vs Phase 2B: Dronabinol and Ethanol vs Phase 2B: Dronabinol and Placebo Ethanol vs Phase 2B: Placebo Dronabinol and Placebo Ethanol; The mean difference in average HbO levels (converted to z-scores) between the pre and post-dose scans for conditions where a participant was dosed with dronabinol (i.e., a main effect for dronabinol dose), estimated via a linear model with with a subject-varying intercept and covariates for (a) overall differences between pre and post-dose scans and (b) visit order; Test type: Superiority; p = 0.94, Regression, Linear — The p-value is adjusted for multiple comparisons using the Benjamini-Hochberg method across the two primary outcome measures and six contrasts. Effects were deemed significant for p<0.05; Estimates for p-values were obtained via a non-parametric resampling approach randomly shuffling condition and refitting the data 10,000 times; Mean Difference (Final Values) = -0.038, 95% CI 2-sided [-0.259 to 0.184], Standard Error of Mean 0.113 — Estimate is the mean difference in average HbO level between pre-dose scans and post-dose scans for dronabinol conditions (positive values denote higher HbO levels for post-dronabinol scans)
Statistical Analysis 2: Comparison: Phase 2A: Placebo Dronabinol Only vs Phase 2B: Dronabinol and Ethanol vs Phase 2B: Placebo Dronabinol and Ethanol vs Phase 2B: Placebo Dronabinol and Placebo Ethanol; The mean difference in average HbO levels (converted to z-scores) between the pre and post-dose scans for conditions where a participant was dosed with ethanol (i.e., a main effect for ethanol dose), estimated via a linear model with with a subject-varying intercept and covariates for (a) overall differences between pre and post-dose scans and (b) visit order; Test type: Superiority; p = 0.94, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.018, 95% CI 2-sided [-0.421 to 0.386], Standard Error of Mean 0.206 — Estimate is the mean difference in average HbO level between pre-dose scans and post-dose scans for ethanol conditions (positive values denote higher HbO levels for post-ethanol scans)
Statistical Analysis 3: Comparison: Phase 2A: Placebo Dronabinol Only vs Phase 2B: Dronabinol and Ethanol vs Phase 2B: Placebo Dronabinol and Placebo Ethanol; The mean difference in average HbO levels (converted to z-scores) between the pre and post-dose scans for conditions where a participant was dosed with both dronabinol and ethanol (i.e., the interaction between dronabinol and ethanol doses), estimated via a linear model with with a subject-varying intercept and covariates for (a) overall differences between pre and post-dose scans and (b) visit order; Test type: Superiority; p = 0.94, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.016, 95% CI 2-sided [-0.535 to 0.568], Standard Error of Mean 0.281 — Estimate is the mean difference in average HbO level between pre-dose scans and post-dose scans for the dronabinol + ethanol condition (positive values denote higher HbO levels for post-dronabinol+ethanol scans)

2. Other Pre Specified Outcome: Change in Concentration of Oxygenated Hemoglobin Between Pre-drug and Post-drug Scans During Resting State.
Description: Subjects completed resting-state fNIRS scans before and after receiving a combination of active dronabinol or placebo dronabinol and active ethanol or placebo ethanol. During the task, the fNIRS device was used to capture concentration of oxygenated hemoglobin to assess prefrontal brain activity.
  Outcomes reflect average change from baseline in HbO concentration over pre-dose scan and average change from baseline in HbO concentration over post-dose scan (expected peak intoxication).
Time Frame: The first resting-state scan session was run before dosing (t ≈ -45min). Drug was administered (t = 0min). The second resting-state scan session was run at the time of expected peak high (t ≈ 90min). Each scan session was six minutes in duration.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Δ mol/L
Arm/Group | Phase 2A: Dronabinol Only | Phase 2A: Placebo Dronabinol Only | Phase 2B: Dronabinol and Ethanol | Phase 2B: Dronabinol and Placebo Ethanol | Phase 2B: Placebo Dronabinol and Ethanol | Phase 2B: Placebo Dronabinol and Placebo Ethanol
Number analyzed (Participants) | 119 | 115 | 30 | 31 | 28 | 34
Δ mol/L
  Predose | -0.00000000056 (0.00000014233) | 0.00000000009 (0.00000011881) | 0.00000000198 (0.00000010153) | 0.00000000021 (0.00000015753) | 0.00000000144 (0.00000017047) | -0.00000000051 (0.00000011795)
  Peak | -0.00000000043 (0.00000010544) | 0.00000000115 (0.00000014174) | 0.00000000025 (0.00000008717) | 0.00000000190 (0.00000013848) | 0.00000000195 (0.00000011273) | -0.00000000014 (0.00000008289)
Statistical Analysis 1: Comparison: Phase 2A: Dronabinol Only vs Phase 2A: Placebo Dronabinol Only vs Phase 2B: Dronabinol and Ethanol vs Phase 2B: Dronabinol and Placebo Ethanol vs Phase 2B: Placebo Dronabinol and Placebo Ethanol; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.94, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.163, 95% CI 2-sided [-0.384 to 0.057], Standard Error of Mean 0.113 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Phase 2A: Placebo Dronabinol Only vs Phase 2B: Dronabinol and Ethanol vs Phase 2B: Placebo Dronabinol and Ethanol vs Phase 2B: Placebo Dronabinol and Placebo Ethanol; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.94, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.176, 95% CI 2-sided [-0.588 to 0.237], Standard Error of Mean 0.210 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Phase 2A: Placebo Dronabinol Only vs Phase 2B: Dronabinol and Ethanol vs Phase 2B: Placebo Dronabinol and Placebo Ethanol; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.94, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.187, 95% CI 2-sided [-0.354 to 0.728], Standard Error of Mean 0.276 — [estimate comment as in outcome 1, analysis 3]

ADVERSE EVENTS:
Time Frame: Participant enrollment to study completion, an average of 3 weeks for Phase 2A and 6 weeks for Phase 2B
Description: Any observed or reported adverse event that occurred during the study visit was recorded and monitored by trained study staff. Additionally, at the beginning of each study visit, participants were asked if there were any changes to their physical or mental health since their last study visit.
Arm/Group | Phase 2A: Dronabinol Only | Phase 2A: Placebo Dronabinol Only | Phase 2B: Dronabinol and Ethanol | Phase 2B: Dronabinol and Placebo Ethanol | Phase 2B: Placebo Dronabinol and Ethanol | Phase 2B: Placebo Dronabinol and Placebo Ethanol
All-Cause Mortality (participants affected / at risk) | 0/128 | 0/126 | 0/39 | 0/39 | 0/32 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/128 | 0/126 | 0/39 | 0/39 | 0/32 | 0/38
Other Adverse Events (participants affected / at risk) | 13/128 | 6/126 | 7/39 | 12/39 | 3/32 | 4/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 2A: Dronabinol Only (N=128) | Phase 2A: Placebo Dronabinol Only (N=126) | Phase 2B: Dronabinol and Ethanol (N=39) | Phase 2B: Dronabinol and Placebo Ethanol (N=39) | Phase 2B: Placebo Dronabinol and Ethanol (N=32) | Phase 2B: Placebo Dronabinol and Placebo Ethanol (N=38)
Anxiety (Psychiatric disorders) | 5 (5) | 2 (2) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Cold (Infections and infestations) | 5 (5) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
After reviewing and updating the study record to appropriately reflect the approved protocol, it was determined that the entry for Study Phase is best represented as N/A, rather than Phase 4, as the purpose of the study is NOT to investigate the safety or efficacy of the drug. This study seeks to use dronabinol only to probe and describe brain physiology. The change from Phase 4 to N/A more accurately and reflects the IRB approved protocol, and the aims of the grant that funds the research.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/17/NCT03655717/Prot_002.pdf
  • Statistical Analysis Plan (2022-04-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT03655717/SAP_003.pdf
  • Informed Consent Form (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT03655717/ICF_004.pdf